CLINICAL TRIAL: NCT03557827
Title: Mechanism of Indocyanine Green-based Photodynamic Therapy for Treating Periodontitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 201701035MIPA
Record Dates: First submitted 2018-03-19; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2017-08

CONDITIONS: Periodontal Diseases
Keywords: periodontitis; photodynamic therapy
MeSH Terms: conditions — Periodontal Diseases; Periodontitis | interventions — Photochemotherapy; Indocyanine Green; Lasers, Semiconductor

STUDY DESIGN:
Intervention Model Description: Split-mouth design. Each quadrant receives different treatment
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and outcome assessor were blinded from the arrangement of the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Sham Comparator): Mechanical debridement by periodontal curets alone
  Interventions: Procedure: Mechanical debridement alone
- Photodynamic Therapy (Active Comparator): Mechanical debridement by periodontal curets and supplement with photodynamic appliance
  Interventions: Drug: Photodynamic Therapy with indocyanine green and diode laser

INTERVENTIONS:
Drug: Photodynamic Therapy with indocyanine green and diode laser — mechanical debridement by periodontal curets plus Indocyanine green solution activated by diode laser. The diode laser is classified as a Class I medical device according to the Directive 93/42/EEC
  Other Names: EmunDo
  Arms: Photodynamic Therapy
Procedure: Mechanical debridement alone — Mechanical debridement by periodontal curets alone
  Arms: control

SUMMARY:
The aim of this study was to investigate the mechanism of indocyanine green photodynamic therapy (PDT) in periodontal therapy. The investigators will recruit 80 participants receiving conventional periodontal disease treatment, or can not fully accept the regular periodontal treatment of adult periodontal disease, photodynamic therapy, and oral periodontal disease of the teeth as the control group, before treatment , Gingival crevicular fluid and dental plaque were collected at 6 weeks, and 6 months after the treatment. The biochemical indexes and strains were analyzed and the data of the participants Term periodontal index.

In this study, indocyanine photodynamic therapy can improve the discomfort of patients with periodontal disease and the periodontal index, the treatment area of the bacteria and the inflammatory response will be significantly decreased, and look forward to this study can establish the indigo cyanine light dynamic teeth Week therapies to provide periodontal patients with more comfortable and effective clinical therapy.

DETAILED DESCRIPTION:
The investigators will recruit 80 adult participants (20 to 80 years old) with periodontal disease who do not receive a regular periodontal course of treatment, or who are unable to receive the regular periodontal treatment completely, using a split-mouth design, meaning that participants are treated with photodynamic therapy of the area for the experimental area, while the mouth corresponding to the location of the area without violations of periodontal disease control area. Participants signed the consent form, the first full-mouth calculus removal and oral hygiene education, and in the experimental area after a week to start photodynamic therapy. The investigators will inject indocyanine in the experimental area, and the wavelength of 810 nm, the energy density of 4.5-9 J / cm2 of the diode laser irradiation; indocyanine and will be cleared after the completion of irradiation, the control area will not For any treatment. After the first treatment, a second, identical treatment will be performed at intervals of 7-10 days. If there is no improvement after 6 weeks, the participant will be treated for the third time.

Participants underwent periodontal examinations in the experimental and control areas at the beginning of the first photodynamic therapy (T0), after six weeks (T1), and six months later (T2), and record the periodontal pocket depth Gingival recession, plaque index and gingivitis index were measured, and the gingival crevicular fluid was obtained by sterilizing the paper needle. The gingival crevicular gingival crevicular gingival crevicular gingival crevicular Fluid, and the use of a periodontal curette to obtain subgingival plaque. The gingival crevicular fluid was quantified using the Periotron 8100 and the concentration of proinflammatory cytokines such as IL-1, IL-10, MMP-8, etc. in the gingival crevicular fluid was analyzed by ELISA kits; DNA was extracted and the periodontal pathogens such as P. gingivalis and T. denticola were detected by Realtime PCR.

In addition, pain assessment was performed with a visual analogue scale at the time of initiation of photodynamic therapy, weekly during the first 6 weeks after initiation of photodynamic therapy, and at 6 months after initiation of treatment . Through these clinical, physiological indicators, as well as the subject experience records, more effective and objective assessment of photodynamic therapy and the establishment of adjuvant therapeutic mechanism.

ELIGIBILITY:
Inclusion

1. 20-80 year-old with their own will and oral cleaning ability
2. Patients who have been diagnosed with periodontitis and have completed a periodontal treatment for at least three months
3. More than one full-mouth periodontal pocket more than 5 mm or more, and a history of repeated inflammation

Exclusion

1. With systemic infection
2. Taking antibiotics within the past 2 weeks
3. Pregnant or lactating
4. Current smoker

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in gingival bleeding index | 6 months
  Measure at four surfaces of tooth

SECONDARY OUTCOMES:
Change in probing depth | 6 months
  Measure at six surfaces of tooth
Change in clinical attachment level | 6 months
  Measure at six surfaces of tooth
Change in plaque index | 6 months
  Measure at four surfaces of tooth
Change in IL-1b | 6 months
  examine the level in the gingival crevicular fluid
Change in gingival crevicular fluid MMP-8 | 6 months
  examine the level in the gingival crevicular fluid
Change in mental status | 6 months
  Visual analogue scale analysis with a score range of 0-10 (0: no discomfort; 10: severe discomfort). Lower score represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Po-Chun Chang Chang, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan